CLINICAL TRIAL: NCT06674239
Title: Determination of the Effect of an Individualized Education Program on Developing Healthy Lifestyle Behaviors and Preventing Postoperative Metabolic Problems in Patients Receiving a Kidney Transplant: A Randomized Controlled Study
Brief Title: Determining the Effect of Individualized Education Program in Kidney Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Ogr. Uyesi Naile, Assistant Prof., Fenerbahce University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FBU/2020-60
Record Dates: First submitted 2024-10-25; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplantation; Healthy Lifestyle Behaviors; Metabolic Problems

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): In the experimental phase of the study, an informed consent form, patient information form, healthy lifestyle behaviors scale, patient follow-up and evaluation form and education booklet were used.
  Patient Information Form: This form was developed by the researchers. Healthy Lifestyle Behaviors Scale: The scale, which measures the health-promoting behaviors associated with the individual's healthy lifestyle, consists of a total of 52 items.
  Patient Follow-up and Evaluation Form: Metabolic value tests are routinely requested in the institution.
  Education Booklet: An education booklet was created based on the literature and the opinions of three experts.
  Data collection method: Individualized education was given to the experimental group. Then, the "Patient Information Form" and the "Healthy Lifestyle Behaviors Scale" were applied as pre-test and post-test. The laboratory values of the patients were examined and recorded in the "Patient Follow-up and Evaluation Form".
  Interventions: Behavioral: Patient Follow-up and Evaluation Form, Patient Information Form Healthy Lifestyle Behaviors Scale Education Booklet
- Observation (No Intervention): Data collection method: Face-to-face interviews were used to inform the patients in the control group about the study and the interview lasted approximately 10-15 minutes. The patients in the control group signed an "informed consent form". The "Patient Information Form" and the "Healthy Lifestyle Behaviors Scale" were applied as pre-test and post-test in the control group. The laboratory values of the patients were examined and recorded in the "Patient Follow-up and Evaluation Form".

INTERVENTIONS:
Behavioral: Patient Follow-up and Evaluation Form, Patient Information Form Healthy Lifestyle Behaviors Scale Education Booklet — In the experimental phase of the study, an informed consent form, patient information form, healthy lifestyle behaviors scale, patient follow-up and evaluation form and education booklet were used.
  Patient Information Form: This form was developed by the researchers. Healthy Lifestyle Behaviors Scale: The scale, which measures the health-promoting behaviors associated with the individual's healthy lifestyle, consists of a total of 52 items.
  Patient Follow-up and Evaluation Form: Metabolic value tests are routinely requested in the institution.
  Education Booklet: An education booklet was created based on the literature and the opinions of three experts.
  Data collection method: Individualized education was given to the experimental group. Then, the "Patient Information Form" and the "Healthy Lifestyle Behaviors Scale" were applied as pre-test and post-test. The laboratory values of the patients were examined and recorded in the "Patient Follow-up and Evaluation Form".
  Arms: Education

SUMMARY:
Objective: The aim of this study is to determine the effect of an individualized education program on the development of healthy lifestyle behaviors and the prevention of postoperative cardiometabolic problems in patients undergoing kidney transplantation. Methods: The study was conducted in the organ transplantation unit of a private hospital between July 2021 and July 2022. The sample size of this randomized controlled trial was determined through power analysis. Patients were randomized into groups using software. Two groups were formed, experimental and control groups, each with 30 patients. Informed consent forms were signed by patients in the experimental and control groups. Data were collected using the "Patient Information Form" and the "Healthy Lifestyle Behaviors Scale" applied as pre-test and post-test. Laboratory values of the patients were examined and recorded in the "Patient Follow-up and Evaluation Form".

DETAILED DESCRIPTION:
Kidney transplantation is the most effective way to reduce high morbidity and mortality in patients with end-stage renal disease. This success has been further enhanced by improvements in immunosuppressive therapy, surgical techniques, and medical care. However, kidney transplantation does not completely reverse the years of decreased renal function and damage caused by dialysis. In addition, new irritants (especially immunosuppressives) added in the post-transplant period can cause problems such as weight gain, impaired glucose tolerance, or diabetes, hypertension, and lipid disorders. Unhealthy lifestyle habits can increase the risk of medical complications in dialysis and transplant patients. On the other hand, the presence of these complications reduces graft efficiency in patients and increases cardiovascular risk. Post-transplant care requires the involvement of multidisciplinary healthcare professionals who must work collaboratively with the patient, the patient's family, and healthcare providers. The outcomes of kidney transplantation are significantly affected by the kidney recipient's ability to adhere to a complex and ongoing self-management regimen. Nurses play an important role in developing the patient's self-efficacy and transforming him/her from a dependent person to a self-sufficient person. The American Nurses Association defines the role of the nurse in health development as "the nurse is responsible for ensuring that individuals and groups adapt to actual and potential health problems, assessing the environment that affects the individual's health, and implementing health-promoting nursing interventions." In this context, the transplant nurse should determine the patient's developmental needs and help him/her acquire healthy lifestyle behaviors, activities of daily living, and preventive practices for self-care. The patient's acquisition of healthy lifestyle behaviors after transplantation should be a part of clinical management. Our literature review showed that studies on this subject are insufficient.

The aim of kidney transplantation is not only to reduce the cost of care while improving kidney function, but also to extend the patient's life, improve the quality of life, and provide a healthy lifestyle and life satisfaction. Considering this information, this study was conducted to determine the effect of an individualized education program on improving healthy lifestyle behaviors and preventing cardiometabolic problems after surgery in kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* patient aged ≥18 years
* literate
* volunteering to participate in the study
* having received a kidney transplant

Exclusion Criteria:

* patient with communication or psychiatric disorder
* having received two or more kidney transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Education given to kidney transplant patients will change healthy lifestyle behaviors. | 1 year
  Healthy Lifestyle Behaviors Scale: Measures the health-promoting behaviors associated with an individual's healthy lifestyle and consists of a total of 52 items and 6 subscales. The lowest score that can be obtained from the scale is 15, and the highest score is 75. As the score obtained from the scale increases, it is seen that the individual has developed a healthy lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Naile Akinci, 1, Principal Investigator — naile.akinci@fbu.edu.tr
Locations (1):
- Fenerbahce University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No